CLINICAL TRIAL: NCT01752101
Title: Identification of a Plasma Proteomic Signature for Lung Cancer
Status: Completed | Type: Observational
Sponsor: Integrated Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: 1013-12
Record Dates: First submitted 2012-11-30; First posted 2012-12-19 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Precancerous Conditions; Carcinoma
Keywords: Precancerous Conditions; Carcinoma
MeSH Terms: conditions — Precancerous Conditions; Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective is to identify a panel of plasma and/or serum proteins that differentiates the absence or presence of lung malignancy in samples obtained from subjects enrolled in this IRB/EC approved study with pulmonary nodules.

DETAILED DESCRIPTION:
Blood samples are obtained from those patients undergoing procedures to determine if a lung nodule is benign or cancerous. The data from the study will not be used to guide or influence the treatment of the patients enrolled in this study. There is no change from the normal standard of care that patients receive.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 40
* any smoking status, e.g. current, former, or never
* co-morbid conditions, e.g. COPD
* Nodule size ≥ 4 mm and ≤ 30 mm (up to Stage 2B eligible), any spiculation or ground glass opacity
* Pathology: malignant - adenocarcinoma, squamous, or large cell
* Pathology: benign - inflammatory (e.g. granulomatous, infectious) or non-inflammatory (e.g. hamartoma)
* Clinical stage, Primary tumor: ≤T2 (e.g. 1A, 1B, 2A and 2B)
* Clinical stage, Regional lymph nodes: N0 or N1 only
* Clinical stage, Distant metastasis: M0 only

Exclusion Criteria:

* prior malignancy within 5 years of lung nodule diagnosis
* No nodule size available
* No pathology data available for those with
* Current diagnosis of non-small cell lung cancer
* Clinical stage: Primary tumor ≥T3; Regional lymph nodes: ≥N2; 4 Distant metastasis: ≥M1

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing procedure for histologic diagnosis of lung nodule(s)
Sampling Method: Probability Sample
Enrollment: 475 (Actual)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Incidence rate of Non-Small Cell Lung Cancer | 24 months after enrollment
  The incidence rate of non-small cell lung cancer in the study population will be correlated to the predictive value of the Sponsor's blood test.

SECONDARY OUTCOMES:
Panel of proteins | At the end of the study
  The positive and negative predictive value of the test to differentiate between malignancy and inflammatory diseases such as granulomatous disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Russell F. Hudnall, Study Director — Integrated Diagnostics, Inc.
Locations (12):
- United States (12):
  - Kaiser Permanente Northern California, San Francisco, California
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - North East Alabama Regional Medical Center, Anniston, Georgia
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Cincinnati, Cincinnati, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Cardiopulmonary Research Science and Technology Institute, Dallas, Texas
  - Intermountain Healthcare, Murray, Utah
  - Group Health Research Institute, Seattle, Washington

REFERENCES:
- [Derived] Kearney P, Hunsucker SW, Li XJ, Porter A, Springmeyer S, Mazzone P. An integrated risk predictor for pulmonary nodules. PLoS One. 2017 May 17;12(5):e0177635. doi: 10.1371/journal.pone.0177635. eCollection 2017. PMID 28545097
- [Derived] Vachani A, Hammoud Z, Springmeyer S, Cohen N, Nguyen D, Williamson C, Starnes S, Hunsucker S, Law S, Li XJ, Porter A, Kearney P. Clinical Utility of a Plasma Protein Classifier for Indeterminate Lung Nodules. Lung. 2015 Dec;193(6):1023-7. doi: 10.1007/s00408-015-9800-0. Epub 2015 Sep 16. PMID 26376647